CLINICAL TRIAL: NCT04080986
Title: DOuble SEquential External Defibrillation for Refractory Ventricular Fibrillation (DOSEVF) Randomized Controlled Trial
Brief Title: DOuble SEquential External Defibrillation for Refractory VF
Acronym: DOSEVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Peel Regional Paramedic Services (Unknown); Toronto Paramedic Services (Unknown); Halton Region Paramedic Services (Other); County of Simcoe Paramedic Services (Unknown); London Health Sciences Centre (Other); Middlesex-London EMS (Unknown); Ottawa Paramedic Service (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DOSEVF RCT
Record Dates: First submitted 2019-08-30; First posted 2019-09-06 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Ventricular Fibrillation
Keywords: Resuscitation; Arrhythmia, Cardiac; Heart Diseases; Heart Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Ventricular Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Heart Arrest

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized trial, with cluster units defined by EMS agency. Each cluster will crossover at six month intervals for each EMS agency during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Arm (No Intervention): All defibrillation attempts will occur using the standard defibrillation method, i.e. defibrillation pads will be placed in the anterior-anterior configuration. The patient may also be administered antiarrythmic agents and epinephrine, as per current provincial standard.
- Double Sequential Defibrillation (Active Comparator): The first three shocks will occur with defibrillation pads placed in the anterior-anterior position. For all further shocks, a second set of defibrillation pads (via a second on scene EMS or fire defibrillator) will be applied in the anterior-posterior position, and defibrillation will be carried out by sequential defibrillation shocks provided by the two defibrillators (i.e. with a short delay between the two defibrillators). The patient may also be administered antiarrythmic agents and epinephrine, as per current provincial standard.
  Interventions: Procedure: Double Sequential Defibrillation
- Vector Change Defibrillation (Active Comparator): The first three shocks will occur with defibrillation pads placed in the anterior-anterior position. All further shocks will occur with the pads placed in the anterior-posterior position. The patient may also be administered antiarrythmic agents and epinephrine, as per current provincial standard.
  Interventions: Procedure: Vector Change Defibrillation

INTERVENTIONS:
Procedure: Double Sequential Defibrillation — Defibrillation using pad placement in anterior-posterior position
  Arms: Double Sequential Defibrillation
Procedure: Vector Change Defibrillation — Defibrillation using two defibrillators, one with pad placement in anterior-posterior position and the other with pad placement in anterior-anterior position delivering two rapid sequential shocks.
  Arms: Vector Change Defibrillation

SUMMARY:
Despite significant advances in resuscitation efforts, there are some patients who remain in refractory ventricular fibrillation (VF) during out-of-hospital cardiac arrest. Double sequential external defibrillation (DSED) and vector change defibrillation have been proposed as viable options for patients in refractory VF. This cluster randomized trial will compare (1) continued resuscitation using standard defibrillation; (2) resuscitation involving DSED; or (3) resuscitation involving vector change defibrillation, in patients presenting with refractory VF during out-of-hospital cardiac arrest. The results of this study will provide high level evidence of the impact of both DSED and vector change defibrillation on ROSC and patient survival after OHCA.

DETAILED DESCRIPTION:
Double sequential external defibrillation (DSED) and vector change defibrillation have been proposed as viable options for patients in refractory ventricular fibrillation (VF) during out-of-hospital cardiac arrest. However, currently there is insufficient evidence to support widespread implementation of this therapy. As such, a well-designed randomized controlled trial (RCT) employing a standardized approach to alternative defibrillation strategies early in the treatment of refractory VF is required to determine whether these treatments may impact clinical outcomes. This cluster randomized trial will be conducted in the regions of Peel, Halton, Simcoe, and the cities of London, Ottawa, and Toronto, Ontario, Canada over a three year time period. All adult (≥ 18 years) patients presenting in refractory VF/pulseless ventricular tachycardia (pVT) (defined as patients presenting in VF/pVT and remaining in VF/pVT after three consecutive standard defibrillation attempts each separated by 2 minutes of CPR) during out-of-hospital cardiac arrest of presumed cardiac etiology will be assigned to be treated by one of three strategies: (1) continued resuscitation using standard defibrillation; (2) resuscitation involving DSED (two defibrillators, one using anterior-posterior pad placement and the second using anterior- anterior pad placement delivering two rapid sequential shocks for all subsequent defibrillation attempts); or (3) resuscitation involving vector change (change of defibrillation pads from anterior-anterior to an anterior-posterior pad position) defibrillation. All study arms will continue to receive antiarrhythmic use and epinephrine as per current provincial standards. The cluster units will be defined by emergency medical service (EMS) agency and each cluster will crossover at 6 month intervals throughout the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Non-traumatic cardiac arrest of presumed cardiac etiology
* Presenting rhythm of ventricular fibrillation or pulseless ventricular tachycardia
* No ROSC or non-shockable rhythm after three consecutive shocks by EMS or fire department.

Exclusion Criteria:

* Traumatic cardiac arrest
* Patients with pre-existing do not resuscitate orders
* Patients without VF or pulseless VT as presenting rhythm
* Patients without three consecutive shocks delivered
* Patients initially treated by non-participating fire or EMS agencies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Survival to Hospital Discharge | Through study completion of three years
  Binary outcome of whether the patient was discharged alive from hospital or died prior to discharge.

SECONDARY OUTCOMES:
Neurologic outcome | Throughout study completion of three years
  Neurologic outcome as defined by the modified Rankin Scale at time of hospital discharge. mRS 0-2 will be considered a good neurologic outcome.
Return of Spontaneous Circulation | 1 Day
  Binary outcome of whether or not a patient had a return of spontaneous circulation
VF termination after first interventional shock | 1 Day
  Cessation of the VF waveform on defibrillator monitor at first rhythm analysis post interventional or standard shock. The interpretation will occur after three standard shocks have failed to terminate VF
VF Termination after all interventional shocks | 1 Day
  Cessation of the VF waveform on defibrillator monitor at any rhythm analysis post interventional or standard shock. The interpretation will occur after three standard shocks have failed to terminate VF
Number of defibrillation attempts to achieve Return of spontaneous circulation | 1 Day
  Total number of shocks required to achieve the first return of spontaneous circulation during resuscitation, inclusive of the first three standard shocks

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Cheskes, MD, Principal Investigator — Sunnybrook Centre for Prehospital Medicine
Locations (6):
- Canada (6):
  - Peel Regional Paramedic Service, Brampton, Ontario
  - Middlesex-London Paramedic Service, London, Ontario
  - Halton Region Paramedic Services, Oakville, Ontario
  - Ottawa Paramedic Service, Ottawa, Ontario
  - County of Simcoe Paramedic Services, Simcoe, Ontario
  - Toronto Paramedic Services, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drennan IR, Dorian P, McLeod S, Pinto R, Scales DC, Turner L, Feldman M, Verbeek PR, Morrison LJ, Cheskes S. DOuble SEquential External Defibrillation for Refractory Ventricular Fibrillation (DOSE VF): study protocol for a randomized controlled trial. Trials. 2020 Nov 26;21(1):977. doi: 10.1186/s13063-020-04904-z. PMID 33243277
- [Background] Cheskes S, Dorian P, Feldman M, McLeod S, Scales DC, Pinto R, Turner L, Morrison LJ, Drennan IR, Verbeek PR. Double sequential external defibrillation for refractory ventricular fibrillation: The DOSE VF pilot randomized controlled trial. Resuscitation. 2020 May;150:178-184. doi: 10.1016/j.resuscitation.2020.02.010. Epub 2020 Feb 19. PMID 32084567
- [Derived] Cheskes S, McLeod SL. Double sequential external defibrillation for refractory ventricular fibrillation: the science, the controversies and the future. J Electrocardiol. 2025 Jul-Aug;91:154046. doi: 10.1016/j.jelectrocard.2025.154046. Epub 2025 Jun 4. PMID 40483934
- [Derived] Cheskes S, Verbeek PR, Drennan IR, McLeod SL, Turner L, Pinto R, Feldman M, Davis M, Vaillancourt C, Morrison LJ, Dorian P, Scales DC. Defibrillation Strategies for Refractory Ventricular Fibrillation. N Engl J Med. 2022 Nov 24;387(21):1947-1956. doi: 10.1056/NEJMoa2207304. Epub 2022 Nov 6. PMID 36342151

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT04080986/Prot_SAP_000.pdf